CLINICAL TRIAL: NCT00730717
Title: Multi Center, Open Label Pilot Study to Determine the Safety and Efficacy of Adalimumab in the Treatment of Pyoderma Gangrenosum
Brief Title: Safety and Efficacy Study of Humira in Treatment of Pyoderma Gangrenosum
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: Stanford University (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Michael Heffernan, MD, Wright State University School of Medicine, Department of Dermatology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM 04-37
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients who are not concurrently receiving methotrexate treatment for pyoderma gangrenosum
  Interventions: Drug: Humira
- 2 (Experimental): Patients who are receiving concurrent methotrexate for pyoderma gangrenosum
  Interventions: Drug: Humira

INTERVENTIONS:
Drug: Humira — Will receive 80 mg of Humira injection at week 0 followed by 40 mg weekly Humira injection from Week 1 to Week 23
  Arms: 1
Drug: Humira — Will receive 40 mg Humira injection every other week from Week 0 to Week 23
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Humira in the treatment of pyoderma gangrenosum.

DETAILED DESCRIPTION:
Pyoderma gangrenosum (PG) is an uncommon dermatosis that consists of nodules and pustules that ulcerate. PG can occur anywhere on the body. Lesions often progress in size and may be multiple. There is no universally accepted treatment for PG. In mild disease, therapy consists of local wound care and topical or intralesional corticosteroids. For more severe disease, systemic agents are necessary. Systemic corticosteroids are often effective, but large doses are required leading to serious long-term side effects. Other immunosuppressives have been reported to be successful in individual case reports and small case series. However, they too are associated with significant toxicities.

Infliximab is an antibody directed against TNF-α. It had been used in success for treatment of PG. Adalimumab (Humira) is a fully human antibody directed against TNF-α. Given that adalimumab has the same target as infliximab, one would expect that adalimumab may also be effective in the treatment of PG. Treatment with adalimumab may be advantageous over infliximab because it can be given at home, whereas infliximab is delivered intravenously in the office. Additionally, because adalimumab is fully human, patients would be less likely to form antibodies against the medication. Purpose of this study is to determine the safety and efficacy of Humira in the treatment of pyoderma gangrenosum.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent.
* Subject is willing and able to participate in the study as an outpatient and is willing to comply with study requirements.
* Subject is 18 years of age or older.
* Subject has a diagnosis of pyoderma gangrenosum that involves total area of 3 cm2 or greater and is of sufficient severity to warrant systemic agents.
* If female of childbearing potential, subject will have a negative urine pregnancy test at Screening and Week 0.
* If female, subject will be either post-menopausal for > 1 year, surgically sterile (hysterectomy or bilateral tubal ligation), or practicing one form of birth control (abstinence, oral contraceptive, estrogen patch, implant contraception, injectable contraception, IUD, diaphragm, condom, sponge, spermicides, or vasectomy of partner). Female subjects will continue to use contraception for 6 months following the last injection.
* Screening laboratory results are within the following parameters:

  * Hemoglobin > 9 g/dL
  * White blood cells > 3.0 x 10 to the 9th power/L, <14.0 x 10 to the 9th power/L (unless on oral corticosteroids and no signs/symptoms of infection)
  * Neutrophils > 1.5 x 10 to the 9th power/L
  * Platelets > 100 x 10 to the 9th power/L
  * Lymphocytes > 0.5 x 10 to the 9th power/L
  * Serum creatinine within 1.5 times the upper limit of normal range
  * AST and ALT within 2 times the upper limit of normal range
  * Subject has been on a stable dose of antibiotics, oral corticosteroids or other immunosuppressives, such cyclosporine, tacrolimus, azathioprine, methotrexate, or mycophenolate mofetil over the previous 4 weeks

Exclusion Criteria:

* Subject has evidence of a clinically significant, unstable or poorly controlled medical condition.
* Subject has a chest X-ray consistent with an active infection or previous exposure to TB and/or a positive purified protein derivative test at screening (>5 mm). (Subjects may participate if they are being actively treated in accordance with CDC guidelines.)
* Subject has a serious, active or recurrent bacterial, viral, or fungal infection. This includes hepatitis B and C, and HIV.
* Subject has been hospitalized for infection or received IV antibiotics within the previous 2 months prior to baseline.
* Subject has clinical evidence as determined by the investigator of acutely infected pyoderma gangrenosum or subject is receiving systemic antibiotics for the treatment of acute infection. Subjects receiving minocycline, tetracycline, dapsone, or other antibiotics for anti-inflammatory purposes are permitted.
* Subject has a history of tuberculosis without documented adequate therapy.
* Subject has a history of a central nervous system disorder/demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis.
* Subject has current signs or symptoms or history of systemic lupus erythematosus.
* Subject has been diagnosed with a malignancy within the past 5 years except for successfully treated non-melanoma skin cancer.
* Subject has signs or symptoms suggestive of a possible lymphoproliferative disease.
* Subject has a diagnosis of severe congestive heart failure (Class III or IV NYHA).
* Subject has had a substance abuse problem within the previous 3 years.
* Subject has been treated with an anti-TNF biologic immune response modifier, such as infliximab, adalimumab, or etanercept within the past 8 weeks.
* Subject has any dermatologic disease in the target site that may be exacerbated by treatment or interfere with examination.
* Subject has been administered an investigational drug in another clinical study within 30 days prior to baseline (or 5 half-lives, whichever is longer).
* Subject has a known allergy to adalimumab.
* Subject is female and is pregnant, is considering becoming pregnant during the study and for 6 months afterwards, or is nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in the number of ulcers from baseline to the end of study | week 0, week 1, week 4 and then very 4 weeks until week 24.
Mean change in ulcer area from baseline to end of study | week 0, week 1, week 4 and then very 4 weeks until week 24.

SECONDARY OUTCOMES:
Number of complete responders, partial responders, minimal responders and non-responders at the end of study. | week 0, week 1, week 4 and then very 4 weeks until week 24.
Mean change in the number of ulcer by visit | week 0, week 1, week 4 and then very 4 weeks until week 24.
Mean change in the ulcer area from baseline by visit | week 0, week 1, week 4 and then very 4 weeks until week 24.
Mean change in subject's evaluation of severity measured by visual analogue scale | week 0, week 1, week 4 and then very 4 weeks until week 24.
Mean change in subject's evaluation of pain by visual analogue scale | week 0, week 1, week 4 and then very 4 weeks until week 24.
Mean change in undermining score | week 0, week 1, week 4 and then very 4 weeks until week 24.
Change in dose of antibiotics and immunosuppressives used to treat PG | week 0, week 1, week 4 and then very 4 weeks until week 24.

CONTACTS AND LOCATIONS:
Overall Officials: David F Fiorentino, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States